CLINICAL TRIAL: NCT06305923
Title: The Efficacy of a Cosmetic Preparation Containing Sheep Colostrum on Mature Skin
Acronym: COLMATSKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RNN/275/21/KE; 503/3-066-02/503-31-001 (Other Grant/Funding Number: Medical University of Lodz)
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Skin Aging
Keywords: sheep colostrum; skin; hydration; TEWL; firmness; mature skin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo cream (Placebo Comparator): everyday using of placebo cream
  Interventions: Other: placebo cream
- colostrum cream (Active Comparator): everyday using of colostrum cream
  Interventions: Other: colostrum cream

INTERVENTIONS:
Other: colostrum cream — the intervention in our study is everyday using a cream with active ingridient
  Arms: colostrum cream
Other: placebo cream — using a placebo cream
  Arms: placebo cream

SUMMARY:
The goal of this clinical trial is to learn about colostrum as a cosmetic in mature skin. . The aim of the study was to examine the effect of a cosmetic preparation containing sheep colostrum on skin with signs of aging in mature women Participants will be given the creams and asked to apply one -two doses in the evening after nighttime facial cleaning. They were also asked to use sunscreens during the day. During the first visit and after eight weeks of everyday use of the tested cream, the skin parameters will be measured three times on both cheeks, and the results were averaged.

Participants will be enrolled to the colostrum cream or base cream groups and will not be informed which group they belonged to.

DETAILED DESCRIPTION:
Participants will be enrolled to the colostrum cream or base cream groups and will not be informed which group they belonged to.

Participants will be given the creams and will be asked to apply one -two doses in the evening after nighttime facial cleaning. They will be also asked to use sunscreens during the day.

1. Instrumental Measurements of Skin Parameters During the first visit and after eight weeks of everyday use of the tested cream, the skin parameters will be measured three times on both cheeks, and the results will be averaged.

   The skin will be measured at standardized temperature and humidity using a Courage + Khazaka electronic GmbH Multi Probe Adapter with the use of the following probes:
   * Corneometer® CM825 probe: measuring skin hydration based on water content in the stratum corneum;
   * Tewameter® TM probe: assessing transepidermal water loss;
   * Mexameter® MX18 probe: measuring the level of hemoglobin (erythema) and mel-anin, the two main dyes responsible for skin color;
   * Sebumeter® SM 815 probe: measuring skin sebum level, independent of water con-tent;
   * Cutometer® MPA 580 probe: measuring the viscoelastic properties of the skin. The R0 and F0 parameters were chosen. R0 represents the passive response of the skin to force, lower values indicate greater firmness. F0 - firmness of the skin at the time of suction. Lower values indicate more elastic skin.
2. Photodocumentation The skin will be subjected to photodocumentation at the first and last visit with the use of the Photomedicus system. The photos will be taken in standard light and with stand-ardized face positions. The photos will be compared using the following scale: 0 means no improvement (the same as the initial picture), 1 - slight improvement, 2 - moderate improvement, 3 - marked improvement (marked improvement in appearance from the initial condition, but not completely optimal), 4 - greatest possible improvement (optimal aesthetic result).
3. Subjective assessment of the skin All participants, i.e. in both groups, subjectively will assess their skin condition after eight weeks of treatment. Participants will rate smoothing of shallow wrinkles, skin tone alignment, regeneration, hydration, elasticity, softness, redness reduction and hypersen-sitivity reduction; they will indicate either improvement, deterioration or no change. Finally, the results in each group will be presented as the percentage of subjects with improved, worsened or unchanged skin.

ELIGIBILITY:
Inclusion Criteria:

* Signs of skin aging: wrinkles, loss of skin elasticity, discolorations, dryness
* Signed informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Allergic to milk proteins
* Suffer from neoplasms, contagious infections, autoimmunologic diseases
* Suffer from face skin diseases
* Have had an aesthetic procedure on the skin of the face during the last two months
* Have been treated with isotretinoin or other oral retinoids during the last six months

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
hydration | 8 weeks
  The skin was measured at standardized temperature and humidity using Courage + Khazaka electronic GmbH Multi Probe Adapter with the use of the aproporate probe.
  Hydratioan - measurement with corneometer, a capacitance method. The results are shown in in arbitrary units between 0 and 130. 1 CU =0,02 mg water in 1 cm2 epidermal stratum corneum
transepidermal water loss | 8 weeks
  The measurement is taken by Tewameter® TM probe: assessing transepidermal water loss. The results are shown in g/h/m2
erythema and melanin content | 8 weeks
  Mexameter® MX18 probe: measuring the level of hemoglobin (erythema) and melanin, the two main dyes responsible for skin color; a broad scale (0-999) of arbitrary Mexameter® units. The Mexameter ® MX 18 probe emits 3 specific light wavelengths. A receiver measures the reflection from the skin. As the quantity of emitted light is defined, the quantity of light absorbed by the skin can be calculated.
sebum | 8 weeks
  Sebumeter® SM 815 probe: measuring skin sebum level, independent of water content; results are shown as Sebumeter® units from 0-350 (approximated to μg/cm 2 in a certain range)

SECONDARY OUTCOMES:
firmness of the skin | 8 weeks
  The skin was measured at standardized temperature and humidity using Courage + Khazaka electronic GmbH Multi Probe Adapter with the use of the following probe: Cutometer® MPA 580 probe: measuring the viscoelastic properties of the skin. R0 represents the passive response of the skin to force, lower values indicate greater firmness. First max. amplitude, highest point of the curve, this has an implication for the firmness of the skin.
  Results in mm. Lower values indicate more elastic skin.
firmness of the skin | 8 weeks
  F0 - firmness of the skin at the time of suction.Area dedicated to the firmness of the skin - the skin deformation under the negative pressure - changes in time - mm*s.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data enclose photos of participants